CLINICAL TRIAL: NCT05037370
Title: Topography-guided vs. Wavefront Optimized Corneal Refractive Surgery: A Prospective Contralateral Randomized Double-masked Study
Brief Title: CONTOURA vs WFO Ablation PRK & LASIK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWH20200077H
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Refractive Surgery
Keywords: Photorefractive Keratectomy (PRK); Laser-assisted in situ Keratomileusis (LASIK); Wave-Front Optimized (WFO); Topography guided ablation

STUDY DESIGN:
Intervention Model Description: Randomized contralateral double-masked study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient will be blinded as to which eye receives which treatment, but the surgical team will not be blinded as to which procedure is performed. Post-operatively, the ophthalmic technicians and optometrists responsible for postoperative examinations will be blinded as to which eye underwent Contoura vs WFO.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LASIK refractive surgery (Experimental): Contralateral Randomize Wave-Front Optimized (WFO) ablation vs Topography-guided ablation
  Interventions: Device: Wave-Front Optimized (WFO) ablation vs Topography-guided (TG) ablation
- PRK refractive surgery (Experimental): Contralateral Randomize Wave-Front Optimized (WFO) ablation vs Topography-guided ablation
  Interventions: Device: Wave-Front Optimized (WFO) ablation vs Topography-guided (TG) ablation

INTERVENTIONS:
Device: Wave-Front Optimized (WFO) ablation vs Topography-guided (TG) ablation — Patient will undergo PRK or LASIK using WFO ablation in one eye and TG ablation on contralateral eye

SUMMARY:
This is a prospective randomized contralateral double-masked study. Each patient will be randomized as to which eye undergoes wave-front optimized (WFO) vs. wave-front guided (WFG) during Photorefractive keratectomy (PRK) or Laser-assisted in situ Keratomileusis (LASIK) surgery to determine which ablation profile provides the best visual outcome.

DETAILED DESCRIPTION:
In 2015, the FDA approved a new laser ablation profile for performing laser corneal refractive surgery. Multiple sophisticated profiles have been developed in an attempt to optimize visual outcomes and reduce post-operative lower and higher-order optical aberrations. Among these include wave-front optimized (WFO) and wave-front guided (WFG) ablation profiles. The former compensated for corneal curvature to reduce spherical aberration and the latter, a more complicated ablation profile, was designed to minimize specific aberrations in an individual eye. Topographic profiles have also been used for over 17 years. These profiles consider the shape of the anterior corneal surface. The newest such topographic ablation profile, Contoura Vision, is a topography guided (TG) profile that, based on over 22,000 curvature data points captured using the VARIO Topolyzer, individualizes the ablation pattern. For comparison, WFO uses a patient's estimated average corneal curvature alone to create an ablation pattern. The addition of the VARIO Topolyzer adds a significant increase of pre-operative patient preparation. Anecdotally, between 1-3hrs of additional technician hours are required to prepare a patient for the Contoura Vision TG ablation profile.

This will be a prospective randomized contralateral double-masked study. Patients will undergo the same standard of care preoperative evaluation and education as any other patient not enrolled in the study. The physician performing surgery will choose either LASIK or PRK, taking into account patient preference, preoperative data and overall clinical picture, ultimately choosing which is best for the patient. If a patient qualifies for both, the patient may choose either LASIK or PRK. Each patient will be randomized as to which eye undergoes a WFO treatment vs Contoura. At the time of surgery the patient will be blinded as to which eye receives which treatment, but the surgical team will not be blinded as to which procedure is performed. Post-operatively, the ophthalmic technicians and optometrists responsible for postoperative examinations (measurement of visual acuity, refractions, transcription of PRO's) will be blinded as to which eye underwent Contoura vs WFO. While treatments will vary, both have the same safety profile. Both involve sophisticated lasers to change the shape of the cornea to achieve the desired outcome. The variance comes in the type of pattern the laser uses to treat each individual. All post-operative care will be standard of care with medications being the same as if the patient were not enrolled in the study. Post-operative evaluations will take place at postoperative day 1, week 1, month 1, month 3, and month 6.

All data collected will be standard pre- and post-operative ophthalmic refractive surgery measurements. This includes a standard medical history, especially to include prior eye surgeries or diseases. Pre-operative measurements include vision assessments, contrast sensitivity, pre- and post-dilation as well as keratometry and axial length measurements. The Contoura requires a separate set of data collection via the VARIO topolyzer. Intraoperative data collected will include variables such as actual treatment outcomes and laser settings. Post-operative measurements will consist of many of the same measurements as those obtained preoperatively including uncorrected and corrected visual acuity, and refractive measurements. A symptoms-based questionnaire specific to corrective eye surgery (PROWL) will be given to patients before and after surgery during routine follow-ups. Each PROWL is specific to an individual eye, not specific to the surgery performed in each eye (i.e. the same PROWL questionnaire will be used regardless of whether the patient underwent PRK or LASIK). All PROWL data will be compared pre- and post-operatively and will be stratified based on surgery.

ELIGIBILITY:
Inclusion Criteria:

* Meet requirements for PRK or LASIK i.e., Stable <= .5 D change MRSE)
* DOD beneficiaries age 21-50 years
* Local pts (w/i 60 mi) who will be in the area for at least 6 months post surgery
* Willing to complete all required follow-up visits

Exclusion Criteria:

* No meeting requirements for PRK or LASIK
* Desiring monovision treatment
* Anisometropia >2D spherical equivalent
* Prior ocular surgeries / trauma / problem
* History of dry eyes
* Hyperopia
* Mixed astigmatism
* Inability to capture VARIO topolyzer scans
* Pregnant (or who plans to be within 6 months after surgery)
* Breastfeeding any time during the study
* History of herpetic disease

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative refractive error | 6 months post-surgery
  The Post-Operative sphere equivalent refractive error for eyes undergoing Wave-Front Optimized (WFO) ablation vs Topography-guided ablation

SECONDARY OUTCOMES:
Post-operative Uncorrected Visual Acuity | 6 months post-surgery
  The Post-Operative visual acuity for eyes undergoing Wave-Front Optimized (WFO) ablation vs Topography-guided ablation

CONTACTS AND LOCATIONS:
Overall Officials: CHARISMA B EVANGELISTA, MD, Principal Investigator — 59th Medical Wing
Locations (1):
- Joint Warfighter Refractive Surgery Center at WHASC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT05037370/ICF_000.pdf